CLINICAL TRIAL: NCT07065591
Title: Anti-Diabetic Drug, Exercise and Healthy Diet for Knee Osteoarthritis With Overweight/Obesity, a Randomized Controlled Trial
Brief Title: Anti-Diabetic Drug, Exercise and Healthy Diet for Knee Osteoarthritis With Overweight/Obesity
Acronym: ADDED
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Lawrence Lau, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW25-051
Record Dates: First submitted 2025-06-29; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: knee osteoarthritis; diet modification; exercise therapy
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Metformin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): This group of patients will receive metformin (max: 500mgx4=2000mg daily). Both groups will start with an initial dose of 500mg daily and the dose will be gradually titrated to 2000mg daily in 6 weeks to allow patients adopting to the gastrointestinal symptoms. Both groups shall be put on metformin or placebo for 6months and then both groups will stop their respective medications and continue on diet modification and exercise therapy only.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): This group of patients will receive placebo. The placebos will be manufactured with Good Manufacturing Practice (GMP) standard such that each placebo pill will look like metformin pill (500mg). Both groups will start with an initial dose of 500mg daily and the dose will be gradually titrated to 2000mg daily in 6 weeks to allow patients adopting to the gastrointestinal symptoms. Both groups shall be put on metformin or placebo for 6months and then both groups will stop their respective medications and continue on diet modification and exercise therapy only.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — The intervention group will receive metformin (max: 500mgx4=2000mg daily). Both groups will start with an initial dose of 500mg daily and the dose will be gradually titrated to 2000mg daily in 6 weeks to allow patients adopting to the gastrointestinal symptoms. Both groups shall be put on metformin or placebo for 6months and then both groups will stop their respective medications and continue on diet modification and exercise therapy only.
  Other Names: Metfomin
  Arms: Intervention group
Other: Placebo — The placebo group will receive placebo. The placebos will be manufactured with Good Manufacturing Practice (GMP) standard such that each placebo pill will look like metformin pill (500mg). Both groups will start with an initial dose of 500mg daily and the dose will be gradually titrated to 2000mg daily in 6 weeks to allow patients adopting to the gastrointestinal symptoms. Both groups shall be put on metformin or placebo for 6months and then both groups will stop their respective medications and continue on diet modification and exercise therapy only.
  Arms: Placebo

SUMMARY:
Obesity is associated with increased pain with knee osteoarthritis and increase progression of knee osteoarthritis while weight loss intervention has been shown to reduce pain and requirement of total knee replacement. In this study, the investigators will assess using diet modification with exercise, and metformin, a common, safe, diabetes mellitus medication that has been in use for 70 years to achieve better weight control to reduce knee pain. This helps the investigators to understand whether the combined treatment can reduce joint pain, reduce body weight and improve symptoms and requirement of total knee replacement.

DETAILED DESCRIPTION:
Unhealthy diet (high fat, sugar) and physical inactivity result in overweight/obesity, which is the major cause of knee osteoarthritis (KOA). KOA further leads to increased intake of comfort food (unhealthy diet) and reduced exercise due to knee pain, forming a vicious cycle. Overweight and obesity are the main risk factors for the major non-communicable diseases (NCDs) like diabetes, etc. which are additional exacerbating factors for KOA. Compared to other NCDs, KOA is more painful and disabling and therefore it commonly leads to early medical consultation for an obese individual. This provides a unique therapeutic opportunity to conduct weight control intervention and lifestyle modification when they are referred for management and waiting for total knee replacement (TKR). Achieving weight control can reduce their subsequent risk of development of other NCDs which lead to increased mortality, and potentially improve their osteoarthritic symptoms, and potentially avoid TKR.

Overweight and Obesity is defined as body mass index (BMI) exceeding 23 and 25 kg/m2 in Hong Kong respectively. Principal applicant (PA) reviewed the BMI of all KOA patients that subsequently had TKR in our hospitals and found the average BMI were 27.72 (2005-2009), 27.78 (2010-2015), and 28.07 (2016-2021) with the number of obese patients increased more than 6 times in 2016-2021 compared to 2005-2009. 73.74% of them were in obese class I and II in 2016- 2021, compared to just 33% of the whole Hong Kong population (same age group) were in these two classes (Based on Department of Health Population Health Survey). Obesity is disproportionally prevalent among KOA patients in Hong Kong with a worsening trend.

Studies and our pilot have found obese KOA patients have more medical comorbidities, with higher prevalence of metabolic syndrome, with more hypertension, dyslipidemia and impaired fasting glucose/diabetes. They are also associated with higher risks of cardiovascular disease, myocardial infarction, and stroke. Obesity is associated with greater pain while waiting for surgery but also with higher chances of developing various perioperative problems, such as surgical site infections, acute kidney injury, increased narcotics consumption, etc. compared to non-obese patients. Therefore, weight loss interventions for KOA are being explored recently to reduce the requirement of TKR, improve the health of KOA subjects, and improve the outcome if TKRs are eventually performed.

Diet modification to achieve weight loss with exercise therapy have been reported reducing KOA pain and improving physical function like walking distance and stair-climb time, compared to control in RCT (ADAPT trial). And it has been showed combining dietary weight loss and exercise can achieve better pain relief and joint loading than either dietary weight loss or exercise alone (Intensive Diet and Exercise for Arthritis (IDEA) trial). Despite these encouraging results, follow-up study at 3.5 years after initial intervention found participants experienced weight regain and reduced pain relief, suggesting difficulty in maintaining long-term weight loss. This matched our published Mendelian Randomization Study which found high BMI contributes to KOA more than effect of dietary intake.

Metformin, an oral anti-diabetic medication, is considered safe, affordable, and well-tolerated. It has been shown to promote weight loss and is a cost-effective option for long-term use on a large scale. Combining metformin with exercise and a balanced diet has been found to be more effective than using metformin alone. Metformin acts on pathways that are also involved in exercise, helping to reduce feelings of hunger and combat obesity. Additionally, metformin has anti-inflammatory and pain-relieving effects that can benefit individuals with osteoarthritis. Moreover, metformin has been shown to enhance muscle quality and reduce the process of muscle aging.

However, current trials using metformin on KOA did not (1) conduct with diet modification nor exercise therapy, (2) assess muscle improvement, (3) assess reduce in TKR, (4) effects of stopping metformin after changes are achieved.

Overall, metformin may accentuate effect of diet modification and exercise as they may be less reliant on comfort food and could perform exercise better (less hunger/pain/body weight and better muscle). This potentially break the vicious cycle of unhealthy diet/physical inactivity- obesity-osteoarthritis.

Trial objectives and Purpose The aim of the study is to determine metformin on top of exercise therapy and diet modification on reducing knee pain (VAS) over 6 months and increasing opt-out preference of joint replacement waiting list.

Hypothesis It is hypothesized that comparing with placebo, metformin will (1) reduce knee pain (primary outcome), (2) reduce body weight and (3) reduce the need of joint replacement.

Study design This is a randomized, double-blinded, placebo-controlled trial in patient with symptomatic knee OA and overweight or obesity, to determine metformin on top of exercise therapy and diet modification on reducing knee pain (VAS) over 6 months and increasing opt-out preference of joint replacement waiting list. Participants will undergo screening and follow-up at an Orthopaedic clinic, receive diet counseling and a structured exercise program, and then be randomly assigned to either metformin or a placebo for 6 months. Subsequently, there will be a 6-month period without medication, during which outcomes will be measured.

Study procedures:

Patients will be screened and followed up in Orthopaedic clinic, completing questionnaires, X-ray, blood glucose level test and blood tests, with blinded research assistants (RA) performing all measurements. Intervention will be started after initial screening confirming eligibility and consent signed.

Intervention:

All participants will undergo a modified Structured Nonsurgical Treatment Programme (SNTP) of Hospital Authority (HA) that references the IDEA trial. In this modified programme, both intervention and control group will receive diet counselling from dietitians with goal of achieving weight loss of 10% baseline body weight and initial diet plan of energy- intake deficit of 800-1000 kcals/day with minimal 1100 kcal for women and 1200 kcal for men and the calorie distribution goal following the Dietary Reference Intakes for Energy and Macronutrients and previous weight loss trials. Their body weight will be monitored during their scheduled nutrition counselling sessions with dietitians. They will also have exercise program with physiotherapists that are facility-based followed by home-based, and the standardized program consisting of an aerobic session (e.g. 15 min aerobic walking), a strength training session (20 min), a second aerobic session (15 min), and a cool-down session (10 min). The strength-training phase is designed to avoid any possible loss of muscle and bone mass resulting from dietary weight loss.

All patient will be prescribed with a standard dose of regular paracetamol and low dose non- steroid anti-inflammatory drugs instructed to be taken on as needed basis as painkillers, same as current normal practice for these patients.

While on diet modification and exercise therapy, patients will be randomly allocated to receive metformin (max: 500mgx4=2000mg daily)(intervention group) or placebos daily (control group). The placebos will be manufactured with Good Manufacturing Practice (GMP) standard such that each placebo pill will look like metformin pill (500mg). Both groups will start with an initial dose of 500mg daily and the dose will be gradually titrated to 2000mg daily in 6 weeks to allow patients adopting to the gastrointestinal symptoms. Both groups shall be put on metformin or placebo for 6months and then both groups will stop their respective medications and continue on diet modification and exercise therapy only. The 6month medication period is based on several factors: Previous trials showing significant weight loss could be achieved by metformin with this timing and further extending the period may not produce much more weight reduction; 3-6months of metformin were showed to reduce arthritis pain; 4months of metformin improved handgrip strength, gait speed, and SPPB (muscle function/sarcopenia parameters); Importantly, a further 6 month period without medication will tell if continuing metformin is needed to maintain its benefit in weight reduction and pain relief. Therefore, this trial the investigators plan for 6months with medication followed by 6months without medication with outcome measurement.

Randomization and blinding:

Patients will be randomized in a 1:1 ratio to either group by computer generated sequence with block randomization. Allocation concealment and double blinding will be performed by: (1) medications being dispensed by centralized pharmacy only; (2) use of an identical placebo tablet, with scheduled gradual titration; (3) both groups will receive diet modification and exercise therapy such that patients, dietitians and physiotherapists will be blinded to group allocation; and (4) measurement by RA blinded to group allocation. Patients and assessors will be blinded to group allocation.

Safety:

Metformin has a well-known good drug safety profile as registered with the Drug Office, Department of Health. The investigators shall outline all potential adverse reactions in informed consent from common ones like nausea, abdominal pain, etc. to rare like lactic acidosis, etc. and these shall be regularly monitored and any of these will be reported to the ethic committee and funding body. They are closely monitored as they will be seen weekly during the 6-week drug titration, monthly clinic/phone follow-up, and assessment at 0, 3, 6, 12 months, as well as regular encounter with physiotherapists and dietitians.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age between 40 and 80 years old, with overweight or obesity (body mass index ≥23 kg/m2) according to Hong Kong Centre for Health Protection definition of overweight and obesity.
* Knee pain for 6+ months with Visual Analogue Scale (VAS) > 40mm/100mm and
* Meet the American College of Rheumatology criteria for knee OA
* OA referred for consideration for joint replacement

Exclusion Criteria:

* Severe radiographic knee OA (Kellgren-Lawrence grade 4) or severe knee pain (VAS>80mm/100 mm) that could not tolerate further conservative management;
* inflammatory arthritis like rheumatoid arthritis, crystal arthritis, etc.
* Preexisting diabetes on antidiabetic drug or drug allergy to metformin.
* Recent knee surgery of the same knee
* Significant bone loss.
* Concomitant neuromuscular diseases affecting lower limb function.
* renal or liver impairment precluding use of metformin.
* VitaminB12 deficiency

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-07-17 (Estimated)

PRIMARY OUTCOMES:
Pain by visual analogue scale | At 0,1.5, 3, 6 and 12 months
  Measure the change in pain level through visual analogue scale (VAS) (0-100mm)

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | At 0,1.5, 3, 6 and 12 months
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) consists of 24 items divided into 3 subscales Pain (5 items), Stiffness (2 items)Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score.
Body weight | At 0,1.5, 3, 6 and 12 months
  Body weight (kg - kilogram) will be measured at each visit.
Knee stiffness | At 0,1.5, 3, 6 and 12 months
  It is measured by knee range measurement
Physical Activity through questionnaire | At 0,1.5, 3, 6 and 12 months
  It is measured by the International Physical Activity Questionnaire short version. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week).
Willingness to proceed TKR immediately | At 0,1.5, 3, 6 and 12 months
  It is measured as proxy of need of TKR.
Physical performance of the muscle - walk | At 0,1.5, 3, 6 and 12 months
  It is measured by 6-metre walk: time to walk 6 metres without deceleration is taken (average of 2 trials is taken, cut-off <1.0m/s).
Physical performance of the muscle - chair stand | At 0,1.5, 3, 6 and 12 months
  It is measured by 5-time chair stand test: time to rise from chair 5 times is recorded (cut-off≥12 seconds).
Physical performance of the muscle - balance | At 0,1.5, 3, 6 and 12 months
  It is measured by Short Physical Performance Battery (SPPB, cut-off<=9). Patients will perform the balance test first, followed by the gait speed test, and finally the chair stand test. Each test will be scored individually, and the total score will be calculated by summing the scores of all three tests. The overall score ranges from 0 to 12, with 12 indicating the best performance.
Muscle strength - Handgrip strength | At 0,1.5, 3, 6 and 12 months
  It is measured by spring-type handgrip dynamometer (JAMAR Hand Dynamometer) with dominant hand in a maximum-effort isometric contraction (cut-off=M: <28 kg, F: <18 kg)
Appendicular skeletal muscle mass (ASM) | At 0,1.5, 3, 6 and 12 months
  It is measured by Bioelectrical impedance analysis (TANITA DC430MA (Tokyo, Japan) with a precision of 0.05 kg. with cut-off=M: <7.0 kg/m2, F: <5.7 kg/m2)
Patient-reported outcome measure questionnaire | At 0,1.5, 3, 6 and 12 months
  It is measured by Sarcopenia and Quality of Life (SarQoL). The final version of the SarQoL® is composed of 55 items translated into 22 questions rated on a 4-point Likert scale. The questionnaire is scored on 100 points. Higher score reflects a higher quality of life.
Kellgren-Lawrence grade | At 0, 6, 12 months
  It is measured at the X-ray, with grade 1, 2, 3 and 4.
Compliance to the study | At every month, up to 1 year
  It is a monthly phone/clinic follow-up to assess pill count for adherence
Blood glucose test. | At baseline, 6 and 12 months
  All patients will be received blood glucose test at baseline for fitness, 6months and 12 months, measured in mmol/L.
Blood test - Complete blood count | At baseline, 6 and 12 months
  Complete blood count in thousand cells per microliter (K/μL).
Blood test - Liver function test | At baseline, 6 and 12 months
  Liver/renal function test, level of alanine transaminase (ALT) and aspartate transaminase (AST).
Blood test - renal function test | At baseline, 6 and 12 months
  Renal function test in Estimated Glomerular Filtration Rate (eGFR).
Blood test - Vitamin B12 | At baseline, 6 and 12 months
  Vitamin B12 in Picograms per milliliter (pg/mL).
Blood test - Calcium phosphate | At baseline, 6 and 12 months
  Calcium phosphate in millimoles per liter (mmol/L).
Blood test - Vitamin D | At baseline, 6 and 12 months
  Vitamin D in nanomoles per liter (nmol/L).
Blood test - Bone profile | At baseline, 6 and 12 months
  Bone profile in millimoles per liter (mmol/L).
Blood test - HbA1c | At baseline, 6 and 12 months
  HbA1c measures the average blood glucose levels over the past 2 to 3 months, expressed in percentage (%). Normal range below 6.4% in Hong Kong.
Blood test - fasting glucose | At baseline, 6 and 12 months
  A fasting blood glucose test measures the blood sugar level after an overnight fast (usually 8-12 hours). Normal is < 6.0mmol/L in Hong Kong.
Blood test - lipids | At baseline, 6 and 12 months
  Cholesterol level in millimoles per litre (mmol/L).

IPD SHARING:
Plan to Share IPD: No
for further patient privacy protection